CLINICAL TRIAL: NCT01693107
Title: The Canadian Atrial Fibrillation Force Contact Ablation Study
Brief Title: Atrial Fibrillation Force Contact Ablation Study
Acronym: CAFCAS
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: Version 20120423
Record Dates: First submitted 2012-09-17; First posted 2012-09-26 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2012-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter Ablation; Electrophysiology; Cardiac Arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Operator Blinded to Contact Force: Physicians performing the ablation will be blinded to the contact force data

SUMMARY:
This study will be divided into two phases. The purpose of the Phase I registry is to assess the current force being used for ablation of symptomatic paroxysmal AF in a wide range of operators in different Canadian centres with the operators being blinded to the contact force data.

In Phase II of the study, operators will have open use of the force contact data. Phase I and II data will be compared in order to assess the efficiency of using the THERMOCOOL® SMARTTOUCH™ catheter.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia affecting over 5% of the population above the age of 65 years. The use of percutaneous catheter ablation for symptomatic management has increased over the last decade. It is well established that AF ablation is superior to anti-arrhythmic drugs for symptomatic recurrence of AF. Despite this, success rates with a single procedure for paroxysmal AF is approximately 80% with the majority of recurrence due to recovery of lesions or "gaps" found at repeat procedures.

In this study, patients with symptomatic paroxysmal atrial fibrillation (AF) will undergo ablation using a newly Health Canada approved catheter with SmartTouch technology that enables the measurement of catheter tip contact force and direction inside the heart. The purpose of Phase I of the study is to assess the current force being used for ablation of symptomatic paroxysmal AF in a wide range of operators in different Canadian centres with the operators being blinded to the contact force data.

The secondary objective will be to assess whether lesion recovery, as assessed in redo procedures, corresponds to contact force measurements. It is hypothesized that gaps found on repeat procedures will correspond to ablation lesions associated with a lower contact force.

In Phase II, operators will have open use of the force contact data. Phase I and II data will be compared in order to assess the efficiency of using the SmartTouch catheter. It is hypothesized that the open use of contact force data will decrease the procedural time and number of lesions to achieve bidirectional pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or greater.
* Patients undergoing first-time pulmonary vein catheter ablation for AF.
* Patients with paroxysmal AF. Paroxysmal AF will be defined as symptomatic episodes of AF lasting less than 7 days or treated with cardioversion(s) within 48 hours of onset.
* At least one episode of AF must have been documented on telemetry, ambulatory monitor, or 12-lead ECG.
* Patients must be able and willing to provide written informed consent to participate in the clinical study.

Exclusion Criteria:

* Patients with a history of any previous ablation for atrial fibrillation.
* Patients with a previous atriotomy scar, ie. Mitral or tricuspid valve replacement or repair, ASD surgery, cardiac transplant.
* Patients with an intracardiac thrombus
* Patients who are or may potentially be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic paroxysmal atrial fibrillation who have failed antiarrhythmic medications and scheduled for a pulmonary vein isolation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Procedural Time | participants will be followed for the duration of hospital stay, an expected average of 36 hours
  Length of time between first ablation and last ablation

SECONDARY OUTCOMES:
Lesion Recovery | up to 1 year
  Localization of recovered gaps
Ablation Time | participants will be followed for the duration of hospital stay, an expected average of 36 hours
  Total time of ablation used during procedure
Number of ablation lesions | participants will be followed for the duration of hospital stay, an expected average of 36 hours
  Total number of ablation lesions to achieve bidirectional block of all 4 pulmonary veins

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leong-Sit, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada